CLINICAL TRIAL: NCT01418001
Title: A Phase IB/II Study of Gemcitabine and Docetaxel in Combination With Pazopanib (Gem/Doce/Pzb) for the Neoadjuvant Treatment of Soft Tissue Sarcoma (STS)
Brief Title: Gemcitabine and Docetaxel in Combination With Pazopanib (Gem/Doce/Pzb) for the Neoadjuvant Treatment of Soft Tissue Sarcoma (STS)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Comprehensive Cancer Network (Network); University of California, Los Angeles (Other); Washington University School of Medicine (Other); Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-104
Record Dates: First submitted 2011-08-15; First posted 2011-08-16 (Estimated); Results first posted 2016-02-17 (Estimated); Last update posted 2018-01-11 (Actual); Status verified 2017-12

CONDITIONS: Sarcoma; Leiomyosarcoma; Malignant Peripheral Nerve Sheath Tumor; Malignant Fibrous; Histiocytoma/Undifferentiated Pleomorphic Sarcoma
Keywords: GEMCITABINE; GW786034 (PAZOPANIB); TAXOTERE (DOCETAXEL); 11-104
MeSH Terms: conditions — Sarcoma; Leiomyosarcoma; Neurofibrosarcoma; Histiocytoma; Histiocytoma, Malignant Fibrous | interventions — pazopanib; Docetaxel

ARMS (1):
- Pazopanib 400 mg QD - Gemcitabine and Docetaxel in Combination (Experimental): This will be a multicenter single arm phase IB/II trial to evaluate the clinical safety and efficacy of gemcitabine/docetaxel and pazopanib in the neoadjuvant treatment of soft tissue sarcoma.
  Interventions: Drug: Pazopanib 400 mg QD - Gemcitabine and Docetaxel in Combination

INTERVENTIONS:
Drug: Pazopanib 400 mg QD - Gemcitabine and Docetaxel in Combination — Patients who meet the eligibility criteria above will be treated with the combination therapy of Gemcitabine, Docetaxel, and Pazopanib for two cycles and subsequently re-evaluated for treatment effect. If no progression of the tumor is seen, patients will continue with two more cycles of treatment (total four cycles). Those patients who have progression of disease will proceed directly to surgical resection.
  Following completion of neoadjuvant treatment, all patients will have definitive surgical resection. Following recovery from surgery, patients will proceed with adjuvant radiation therapy. Patients will then be followed for 2 years or until January 1st 2015, whichever comes first .

SUMMARY:
The purpose of this study is to see the effects, good and/or bad, of the drug combination of gemcitabine, docetaxel and pazopanib on sarcoma. This is a phase Ib-phase II clinical trial. The goal of a phase Ib part of the clinical trial is to confirm a dose of the drugs that is safe. The investigators determine this by closely checking for side effects that the patient may experience.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed extremity only, ≥8 cm, high grade STS (MPNST, MFH/UPS, LMS) at MSKCC or locally for participating sites.
* Subjects must have only localized disease that is potentially amenable to definitive resection.
* The first 15 MSKCC patients on the Phase II portion of the protocol must undergo either an open incisional or core tumor biopsy prior to the initiation of therapy.
* Patients must have measurable disease by RECIST 1.1, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques or as >10 mm with spiral CT scan. See Section 10 for the evaluation of measurable disease.
* Age >18 years. ECOG performance status 0 or 1.
* Patients must have normal organ and marrow function as defined below (ULN indicates institutional upper limit of normal): Absolute neutrophil count (ANC) ≥1.5 X 109/L Hemoglobin ≥9 g/dL (5.6 mmol/L) Platelets ≥100 X 109/L International normalized ratio (INR) ≤1.2 X ULN Activated partial thromboplastin time (aPTT)≤1.2 X ULN Total bilirubin ≤1.5 X ULN Alanine amino, transferase (ALT) and Aspartate aminotransferase (AST) ≤2.5 X ULN Serum creatinine ≤1.5 mg/dL (133 μmol/L) Or, if serum creatinine, >1.5 mg/dL: Calculated creatinine clearance (ClCR)

  ≥30 mL/min to ≥50 mL/min Urine Protein to Creatinine Ratio (UPC; appropriate appendix) <1 Or, 24-hour urine protein <1g
* Patients must not have current evidence of another malignancy.
* Pazopanib, gemcitabine and docetaxel all carry category D (positive evidence of risk) pregnancy status. For this reason women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) during therapy and for at least 8 weeks after completion of therapy and have pregnancy testing prior to study entry and after two cycles of treatment. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.

Exclusion Criteria:

* Patients who have had major surgery 4 weeks prior to entering the study, or those who have not recovered from adverse events to ≤ NCI CTC AE Grade 1, associated with surgery. Excluded from such considerations are surgical changes not expected to improve, e.g. removal of muscle tissue.
* Patients must not have had been treated previously with radiation, chemotherapy or other anti-cancer agent for the current disease.
* History of allergic reactions or hypersensitivity reactions attributed to compounds of similar chemical or biologic composition to pazopanib, gemcitabine, docetaxel or other agents used in the study.
* Patients with a contraindication to MRIs.
* Patients who required concomitant treatment with medications that are known to be inhibitors or strong inducers of isoenzyme CYP3A4, CYP2C8, and CYP2D6 unless the drugs are medically necessary and no substitutes are available. If there are no acceptable substitutes, special precautions should be taken in these patients. Similarly, co-administration with CYP3A inhibitors (e.g. Ergot derivatives, Neuroleptics, Antiarrhythmics, Immune modulators and miscellaneous agents such quetiapine, risperidone, clozapine, atomoxetine, and inducers (e.g. Glucocorticoids, Anticonvulsants, HIV antivirals, Antibiotics, miscellaneous agents such as St. John's Wort, modafinil, pioglitazone, troglitazone, simvastatin, should also be avoided if possible, or otherwise subject to caution (e.g. increased frequency of safety monitoring). Strong CYP3A4 inhibitors are PROHIBITED within 14 days prior to the first dose of pazopanib including: Antibiotics, HIV protease inhibitors, Antifungals and Antidepressants
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, including HIV, active hepatitis B or C, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, poorly controlled diabetes or psychiatric illness/social situations that would limit compliance with study requirements. Hepatitis B and C will be screened for in all patients prior to initiating treatment via hepatitis B serologic markers, that is, HBsAg, HBs Ab, HBc Ab and Hep C Antibody. If patients have positive serologic markers, viral load markers (HBV-DNA and Hepatitis C RNA-PCR) will be performed during screening to confirm disease as well as screening for hepatitis C via quantitative RNA-PCR.
* Pregnant women and women who are breast-feeding.
* HIV -positive patients on combination antiretroviral therapy due to the potential for pharmacokinetic interactions with pazopanib.
* Patients with significant respiratory compromise or an active and unexplained pneumonitis given that these patients would have an increased risk of pneumonitis from gemcitabine, and would also confuse the evaluation of pneumonitis on the trial
* Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding including, but not limited to:

Active peptic ulcer disease

* Inflammatory bowel disease (e.g. ulcerative colitis, Crohn's disease), or other gastrointestinal conditions with increased risk of perforation
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal
* abscess within 28 days prior to beginning study treatment Active diarrhea of any grade
* Clinically significant gastrointestinal abnormalities that may affect absorption of investigational product including, but not limited to:
* Malabsorption syndrome
* Major resection of the stomach or small bowel
* History of any one or more of the following cardiovascular conditions within the past 6 months:

Cardiac angioplasty or stenting Myocardial infarction Unstable angina Coronary artery bypass graft surgery Symptomatic peripheral vascular disease

* History of cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months.
* Note: Subjects with recent DVT who have been treated with therapeutic anticoagulating agents for at least 6 weeks are eligible
* Corrected QT interval (QTc) ≥ 450 msecs using Bazett's formula (append formula); for subjects with bundle branch block (BBB), QTc ≥480 msecs using Bazett's formula.)
* Poorly controlled hypertension, defined as systolic blood pressure (SBP) of ≥140 mmHg or diastolic blood pressure (DBP) of ≥ 90mmHg.
* Note: Initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry.

History of Class III or IV congestive heart failure, as defined by the New York Heart Association Classification of Congestive Heart Failure [see Appendix D for description]

* Evidence of active bleeding or bleeding diathesis
* Administration of any non-oncologic investigational drug within 30 days or 5 half lives whichever is longer prior to receiving the first dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-08; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Tap, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - UCLA, Los Angeles, California
  - Northwestern University, Evanston, Illinois
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan-Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Pazopanib 400 mg QD: Pazopanib 400 mg QD - Gemcitabine and Docetaxel in Combination with Pazopanib
Period: Overall Study
Arm/Group | Pazopanib 400 mg QD
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Level 1: Pazopanib 400 mg QD Gemcitabine and Docetaxel in Com: Level 1: Pazopanib 400 mg QD - Gemcitabine and Docetaxel in Combination with Pazopanib
Arm/Group | Level 1: Pazopanib 400 mg QD Gemcitabine and Docetaxel in Com
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Overall Objective Response
Description: Overall objective response measured using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: Every 6 weeks up to 2 years
Measure: Number; unit: participants
Groups:
- Level 1: Pazopanib 400 mg QD: Level 1: Pazopanib 400 mg QD - Gemcitabine and Docetaxel in Combination with Pazopanib
Arm/Group | Level 1: Pazopanib 400 mg QD
Number analyzed (Participants) | 5
participants
  Complete Response (CR) | 3
  Stable Disease (SD) | 2

2. Secondary Outcome: Pathologic Response
Description: will be assessed by both MRI and by pathologic review after surgery. An estimate of each response rate and the 95% CI will be provided
Time Frame: 2 years
Population: No data is available because data was not collected due to lack of accrual.
Arm/Group | Pazopanib 400 mg QD
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Level 1: Pazopanib 400 mg QD
Serious Adverse Events (participants affected / at risk) | 3/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Level 1: Pazopanib 400 mg QD (N=5)
Wound infection (Infections and infestations) | 1
Fatigue (General disorders) | 1
Alanine aminotransferase increased (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Level 1: Pazopanib 400 mg QD (N=5)
Alanine aminotransferase increased (Blood and lymphatic system disorders) | 2
Anemia (Blood and lymphatic system disorders) | 4
Aspartate aminotransferase increased (Blood and lymphatic system disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 2
Hoarseness (General disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hypertension (Cardiac disorders) | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 1
Lymphocyte count decreased (Blood and lymphatic system disorders) | 2
Mucositis oral (General disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Platelet count decreased (Blood and lymphatic system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes